CLINICAL TRIAL: NCT02602834
Title: Changes in Blood Measured Before, During and After Exercise in Heart Transplant Recipients. Imminently Effect of Interval Training With High Intensity Compared With Continuous Moderate Intensity
Brief Title: Imminently Effect of Interval Training With High Intensity (HIT) After Heart Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Health Association (Other)
Responsible Party: Principal Investigator, Marianne Yardley, MD, PhD candidate, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2015/97/REK sør-øst A
Record Dates: First submitted 2015-10-06; First posted 2015-11-11 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Heart Transplantation
Keywords: exercise test; biological markers
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HTx (Experimental): Heart transplant recipients n=15
  Interventions: Other: interval training; Other: moderate exercise
- Control (Active Comparator): Healthy controls n=5
  Interventions: Other: interval training; Other: moderate exercise

INTERVENTIONS:
Other: interval training — 4 intervals with high intensity on treadmill, and approximately 3 minutes rest between intervals.
Other: moderate exercise — 30 minutes (moderate intensity) aerobic exercise on treadmill without rest.

SUMMARY:
High intensity Interval training (HIT) has repeatedly been documented to have superior positive effects on oxygen uptake and general physical health compared to continuous moderate exercise in healthy individuals and patients with heart disease. Recently, the same effect has been shown in heart transplanted recipients. Which mechanisms that explains this difference is uncertain; the effect can be due to changes in the heart or changes in the peripheral tissue and muscles. To explore these mechanisms the investigators will in this study compare two different exercise modalities, and explore how different biomarkers change in blood, related to exercise.

DETAILED DESCRIPTION:
15 heart transplanted recipients (and 5 healthy controls) will be included in the study. Each patient will have three study-days.

The study is designed to be a cross-over study. And randomisation will decide which training they will have som training session 1 and training session 2; Interval or continuous training.

Before starting the two training sessions they will measure oxygen uptake and baseline blood samples.

During each exercise session the patients will take blood samples during and after exercise.

After first study admission the patients will have a wash out period for 1 week until first training session, and another week until the last session.

ELIGIBILITY:
Inclusion Criteria (HTx):

* 1-10 years after heart transplantation
* Lives in Oslo or near Oslo
* Stable health condition
* Optimal medical treatment/ medication
* No limiting physical handicap
* Written consent

Inclusion healthy control:

* No verified heart disease
* Willing to preform the study
* Over 18 years
* Written consent

Exclusion Criteria:

* Under 1 year or over 10 year since HTx.
* Lives far from Oslo
* Unstable health condition
* Not optimal medical treatment and/ or medication
* Limiting physical handicap
* Under 18 years
* Not written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Changes in crp with interval training compared to moderate training | 1 week
Changes in interleukin levels with interval training compared to moderate training | 1 week
Changes in ICAM levels with interval training compared to moderate training | 1 week
Changes in MiRNA levels with interval training compared to moderate training | 1 week

SECONDARY OUTCOMES:
Questionnaire of quality of life | baseline
Oxygen uptake | baseline
  V02 peak measured på exercise test on treadmill.
Questionnaire of physical activity | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lars LG Gullestad, professor, Study Director — OUS-Oslo university hospital rikshospitalet, cardiology department
Locations (1):
- OUS- Rikshospitalet, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Yardley M, Ueland T, Aukrust P, Michelsen A, Bjorkelund E, Gullestad L, Nytroen K. Immediate response in markers of inflammation and angiogenesis during exercise: a randomised cross-over study in heart transplant recipients. Open Heart. 2017 Nov 28;4(2):e000635. doi: 10.1136/openhrt-2017-000635. eCollection 2017. PMID 29225901